CLINICAL TRIAL: NCT01001598
Title: Phase I/II Dose Escalation Trial of Danazol in Patients With Fanconi Anemia or Dyskeratosis Congenita
Brief Title: Safety and Efficacy Trial of Danazol in Patients With Fanconi Anemia or Dyskeratosis Congenita
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to under enrollment
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Colin Sieff, Director, Bone Marrow Failure Service, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-03-0131
Record Dates: First submitted 2009-10-22; First posted 2009-10-26 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-01

CONDITIONS: Fanconi Anemia; Dyskeratosis Congenita
MeSH Terms: conditions — Fanconi Anemia; Dyskeratosis Congenita | interventions — Danazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- danazol (Other): Subjects with either Fanconi anemia or Dyskeratosis congenita
  Interventions: Drug: danazol

INTERVENTIONS:
Drug: danazol — Dosage is done according to weight; capsules are 50, 100, 200 mg
  Other Names: Danocrine, Danol, Danatrol

SUMMARY:
Fanconi anemia (FA) and Dyskeratosis congenita (DC) are inherited bone marrow failure syndromes. The current androgen treatments (e.g., oxymetholone) used to treat FA and DC can cause unwanted masculinizing side effects, indicating a need for a different medication. Danazol is a less potent androgen,and may therefore have fewer masculinizing side effects. Danazol is currently approved by the Food and Drug Administration (FDA) for the treatment of other diseases, but it has never been studied in patients with FA and DC.

The main purpose of this study is to see if danazol is a safe treatment for FA and DC. Specifically,we would like to determine:

* the best dose of danazol;
* how fast hemoglobin (a protein that carries oxygen in the blood) levels rise in FA and DC patients receiving danazol therapy; and
* the genetic pattern (known as expression profile) of certain cells in response to danazol, which can predict how well people respond to the medication.

Subjects who enroll in the study will be treated with danazol for up to 24 weeks (about 6 months), and will have up to 11 study visits, including followup visits at 38 weeks (9 months) and 52 weeks (one year).

DETAILED DESCRIPTION:
Eligible patients with either Fanconi anemia (FA) or Dyskeratosis congenita (DC) will initially receive danazol at a dose of 5 mg/kg/d orally, rounded to the nearest 100 mg. For the first 8 weeks, the patient will be evaluated at weeks 2, 5, and 8 for hematologic response (HR). If the patient shows a hematological response (either a hemoglobin or platelet value no longer meeting blood cell count criteria for protocol inclusion in the absence of recent transfusions)within the first 12 weeks on the initial dose, the study drug will be continued at this dose for the next 6 weeks. If the patient fails to show any hematologic response within the first 12 weeks, the dose will be escalated to 10 mg/kg/day for the next 6 weeks, and an additional monitoring visit will be required at week 14. If at week 18, the patient fails to show any hematological response on the increased dose, the dose will be increased to 15 mg/kg/day for another 6 weeks (not to exceed 800 mg/day), and an additional monitoring visit will be required at week 20. At 24 weeks, if there is no response to this dose the patient will be taken off study drug and classified as a treatment failure, and will be monitored at weeks 38 and week 52). After week 24, if the patient continues to show a response, however, the study drug may be continued at the discretion of their primary care physician, with monitoring at weeks 38 and 52.

Should the patient lose the hematologic response on 5 or 10 mg/kg/day dosing at any point within the first 18 weeks of treatment, the dose will be escalated to 10 or 15 mg/kg/day (not to exceed 800 mg/day), respectively. The patient will continue to be evaluated at the next visit. If after week 24 no hematologic improvement is seen, the patient is then taken off study drug and monitored at weeks 38 and 52.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be diagnosed with FA that is documented by a positive test for increased chromosomal breakage with mitomycin C or diepoxybutane. DC patients must have clinical features consistent with the diagnosis, abnormally short lymphocyte telomeres < 1st centile by flow-FISH evaluation, or mutation in one of the known DC genes (DKC1, TERT, TERC, TINF2, NOP10, NHP2).
2. At least the following peripheral blood cytopenias: (without transfusion) Absolute neutrophil count < 500/uL or Platelet count < 30,000/uL or Hemoglobin < 8.0 gm/dl
3. Negative pregnancy test by hCG testing, if of child-bearing potential.
4. Agreement to use a medically approved form of birth control, if of child-bearing potential.
5. Signed informed consent by the patient or legally authorized representative.
6. Patients must be either 3 years of age or > 14 kg.

Exclusion Criteria:

1. Malignancy
2. Concurrent enrollment in any other study using an investigational drug.
3. Concurrent use of anticoagulants.
4. Use of androgen therapy within last three months.
5. Patients with liver disease as defined by SGOT, SGPT or bilirubin greater than the upper limit of normal.
6. Patients with renal disease as defined by serum creatinine greater than the upper limit of normal for age.
7. Patients less than either 3 years of age or 14 kg.
8. Patients who have HLA matched sibling donors.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin A Sieff, MB.BCh, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from clinic and by letter to Pediatric Hematologists in USA
Pre-assignment Details: 1. Patients with documented Fanconi anemia (FA) or dyskeratosis congenita (DC)
  2. Peripheral blood cytopenias (without transfusion, and at least one result obtained in the past two months that meet criteria): ANC < 500/uL or platelets < 30,000/uL or Hb < 8.0 gm/dl
  3. . Not pregnant
  4. Not on birth control
  5. Consent
  6. 3 yrs/ > 14 kg.
Groups:
- Danazol: Subjects with either Fanconi anemia or Dyskeratosis congenita enter a single arm 24 week danazol dose escalation study: Dosage 5mg/kg/d; if no response at 12 weeks increase to 10 mg/kg/d; if no response at 18 weeks increase to 15 mg/kg/d. If no response stop at 24 weeks. Responders continue danazol at discretion of PCP.
Period: Overall Study
Arm/Group | Danazol
Started (Monitoring visits at 2, 5, 8, 12, 18, 24 wks - visits at 14 and/or 20 weeks if dose escalation) | 5
Completed | 3 (3 completed study (2 FA and 1 DC) in 2011)
Not Completed | 2
Not completed — Hematopoietic Stem Cell Transplant | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Danazol
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Toxicity Associated With Danazol Therapy: Virilization, and/or New or Progressive Evidence of Either Hepatic or Renal Toxicity at a Grade II Level Using National Cancer Institute Common Toxicity Criteria (NCI-CTC).
Description: All toxicities were collected and adjudicated to definitely-related, possibly-related, or unrelated to the treatment.
Time Frame: 48 weeks (24 weeks treatment and 24 weeks extension phase)
Population: 4 patients with Fanconi anemia and 1 with dyskeratosis congenita
Measure: Count of Participants; unit: Participants
Arm/Group | Danazol
Number analyzed (Participants) | 5
Participants
  Virilization - definitely related | 2
  Hepatic - possibly related | 1

2. Secondary Outcome: The Optimal Dose and Number of Participants With Hematologic Response Rate in Fanconi Anemia (FA) and Dyskeratosis Congenita (DC) Patients Receiving Danazol Therapy
Description: The optimal dose could not be calculated because the number of participants needed to do this were not enrolled. Hematologic response rate (HR) was calculated for each participant at Week 12, 18, and 24. HR was defined by hemoglobin (Hg), platelets or neutrophil response. Please find the evaluation criteria used below:
  Hemoglobin response: Hgb≥8 g/dL if baseline Hgb≤7 g/dL, or Hgb rise ≥1 g/dL from baseline if baseline Hgb>7 g/dL. No RBC transfusion during the 8 weeks prior to response evaluation.
  Platelet response: Platelet count ≥30,000/ μL if baseline platelet count ≤20,000/ μL, or platelet count rise >10,000/ μL from baseline if baseline platelet count >20,000/ μL. No platelet transfusion during the 4 weeks prior to response evaluation.
  ANC response: ANC count ≥1,000/ μL if baseline ANC count ≤500/ μL, or ANC count rise >500/ μL from baseline if baseline ANC count >500/ μL.
Time Frame: 12, 18 and 24 weeks
Population: 2 participants withdrew before HR could be assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Danazol
Number analyzed (Participants) | 3
Participants
  HR by hemoglobin at 12 weeks | 3
  HR by hemoglobin at 18 weeks | 3
  HR by hemoglobin at 24 weeks | 3
  HR by platelets at 12 weeks | 0
  HR by platelets at 18 weeks | 0
  HR by platelets at 24 weeks | 2
  HR by neutrophils at 12 weeks | 0
  HR by neutrophils at 18 weeks | 0
  HR by neutrophils at 24 weeks | 2

3. Secondary Outcome: The Gene Expression Profile of Progenitor Cells in Response to Danazol, Both to Predict Responsiveness and to Screen for Small Molecules That Show a Profile Similar to That of Responsive Patients
Description: The gene expression profiles were planned to be run on bone marrow samples collected from patients at baseline and 24 weeks but bone marrow was never collected at 24 weeks.
Time Frame: Baseline and 24 weeks
Population: Baseline samples were too noisy to determine gene expression.
Arm/Group | Danazol
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Single Arm Phase I/II Study
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Phase I/II Study (N=5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Danazol started at 5 mg/kg/day (200 mg/day); day 9 a rash that on her hands and spread to the rest of her body diagnosed as hives. Also on birth control (Altavera). Dermatologist at BCH recommended against re-starting the danazol.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Phase I/II Study (N=5)
Mood changes (Nervous system disorders) | 1 (1) — Probably related
Constipation (Gastrointestinal disorders) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) — Enlargement of the left lobe
Virilization (Endocrine disorders) | 2 (2) — Clitoral and phallic enlargement

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No